CLINICAL TRIAL: NCT02989688
Title: Glycaemic Response to Oral Nutrition Support During Haemodialysis
Acronym: GRO-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KingCHL
Record Dates: First submitted 2016-01-20; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes; Chronic Kidney Disease; End Stage Renal Failure on Dialysis
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- modified carbohydrate drink (Active Comparator): Dietary Supplement - renal specific slow release carbohydrate ONS (220 ml Nepro HP (Abbott Nutrition)
  Interventions: Dietary Supplement: Nepro HP (Abbott Nutrition)
- macronutrient matched drink (Active Comparator): Dietary Supplement - 125 ml Fortisip Compact Protein (Nutricia) plus 20ml Calogen (Nutricia)
  Interventions: Dietary Supplement: Fortisip compact protein 125 ml + Calogen 20ml (Nutricia)
- standard drink (Active Comparator): Dietary Supplement - 125 ml Fortisip compact (Nutricia)
  Interventions: Dietary Supplement: Fortisip compact 125 ml (Nutricia)

INTERVENTIONS:
Dietary Supplement: Nepro HP (Abbott Nutrition) — oral nutritional supplement drink with modified carbohydrate composition
  Arms: modified carbohydrate drink
Dietary Supplement: Fortisip compact protein 125 ml + Calogen 20ml (Nutricia) — Fortisip compact protein 125 ml + Calogen 20ml (Nutricia) oral nutritional supplement drink macronutrient matched with standard carbohydrate composition
  Arms: macronutrient matched drink
Dietary Supplement: Fortisip compact 125 ml (Nutricia) — Fortisip compact 125 ml (Nutricia) oral nutritional supplement drink - standard
  Arms: standard drink

SUMMARY:
Patients with kidney, or renal, failure require life-saving treatment with regular dialysis. Dialysis is a form of treatment that simulates some kidney functions; to remove harmful waste products and extra water from the blood. Almost one-third of people with kidney failure also have diabetes, as diabetes is one of the leading causes of kidney disease in the United Kingdom, usually due to poor blood sugar control over a long period of time. Malnutrition is common in patients needing dialysis due to kidney failure causing fatigue, taste changes and a build up of waste products, which can reduce appetite. Treatment of malnutrition involves increasing both the energy and protein intake from food and drinks, and milk-drink style specialist nutrition drinks are often given to dialysis patients due to their specific dietary needs. These nutrition drinks can increase blood sugar levels and optimal control for diabetes may be difficult. This research study aims to measure the blood sugar response to a "slow-release" sugar nutrition drink specifically designed for dialysis patients, which may result in a lower blood sugar level, compared to standard nutrition drinks, consumed during a dialysis session. 28 patients with diabetes and having regular dialysis treatment will enrol in the study. Patients will be asked to drink 1 of 3 different nutrition drinks, once a week for 3 weeks during their regular dialysis treatment. Blood sugar levels will be measured from the blood samples taken from the patient's circulation directly before it enters the dialysis machine over 3 hours and the maximum blood sugar reading and total blood sugar response will be measured. Differences between the 3 drinks will be tested statistically. The results will help to advise patients with diabetes and kidney failure on the most suitable type of nutrition drink to consume during dialysis.

DETAILED DESCRIPTION:
Patients with end stage kidney disease requiring dialysis are at the highest risk for cardiovascular disease, and many of our dialysis population also have diabetes. Malnutrition is common in patients undergoing dialysis and causes are multifactorial. Oral nutrition support is the first line treatment for malnutrition, and often includes the use of liquid nutrition supplements, especially in dialysis patients due to the already restricted diet required to maintain electrolyte balance. Oral nutrition supplements (ONS) can raise serum blood glucose levels and optimal control for diabetes may be difficult when ONS are required. This study aims to evaluate the post-prandial response to a newly re-formulated slow release carbohydrate renal specific oral nutrition supplement, compared to standard and macro-nutrient matched ONS products, during haemodialysis, using a randomised cross-over trial design. 28 patients with diabetes and end stage kidney disease undergoing haemodialysis will be recruited to the study, including 8 in the pilot phase and 20 in the study. Patients will be randomised in a crossover design to 3 study treatments over 3 weeks - slow release CHO ONS, macronutrient matched ONS, and standard ONS. Central blood glucose levels will be measured over 3 hours and the peak and mean incremental area under the curve (iAUC) of the post prandial blood glucose response will be calculated for each study treatment. Differences between treatments will be determined with repeated measures analysis of co-variance (ANCOVA). The acute effect of different nutritional supplements on blood glucose will be discussed in the context of maintaining optimal blood glucose control during dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes
* End stage kidney disease on haemodialysis
* Body mass index 18.5-35kg/m2
* Able to provide written informed consent

Exclusion Criteria:

• Infection or course of antibiotics in the last month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose response curve | 3 hour
  Mean incremental area under the curve for blood glucose response to intervention over 3 hours

SECONDARY OUTCOMES:
Peak blood glucose reading within 3 hours | 3 hours
Appetite score pre and post ONS | 3 hours
  likert scale
Flavour acceptability scale for ONS product | 3 hours
  likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Helen L MacLaughlin, PhD, Principal Investigator — Clinical Lecturer
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133